CLINICAL TRIAL: NCT04266600
Title: Extended Mesenteric Excision in Ileocolic Resections for Crohn's Disease: A Multicenter Prospective Cohort Study
Brief Title: Extended Mesenteric Excision in Ileocolic Resections for Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: Montreal General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Associate Professor of Surgery, Jewish General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MUHC-2020-5789
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Crohn Disease; Recurrence; Crohn's Ileocolitis
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective arm (extended mesenteric resection) (Experimental): Surgery can be performed either laparoscopically or open depending on surgeon preference and the circumstances of the surgery. Surgeons will perform a high ligation of the ileocolic pedicle, between the superior mesenteric artery and the bifurcation of the ileal and right colic branches, and to fully mobilize the mesentery off of the retroperitoneum prior to bowel transection and anastomosis. The entire mesentery related to the specimen will be removed.
  Outcomes in the prospective arm will be compared to historical controls.
  Interventions: Procedure: Extensive mesentery resection
- Retrospective arm (No Intervention): Retrospective patient data will be obtained by querying the Opera operating room database of both study institutions. Electronic records will be analyzed for all patients undergoing a first-time ileocolic resection for Crohn's Disease between January 1, 2009 - December 31, 2018.

INTERVENTIONS:
Procedure: Extensive mesentery resection — Surgeons will perform a high ligation of the ileocolic pedicle, between the superior mesenteric artery and the bifurcation of the ileal and right colic branches, and to fully mobilize the mesentery off of the retroperitoneum prior to bowel transection and anastomosis
  Arms: Prospective arm (extended mesenteric resection)

SUMMARY:
The study is looking at the role of the mesentery in disease recurrence for ileocolic Crohn's disease. It is a prospective study that has been designed to perform extended mesenteric excision on patients undergoing their first ileocolic resection for Crohn's disease. Endoscopic recurrence will be monitored with the hypothesis that patients receiving extended mesenteric ileocolic resection will have reduced endoscopic recurrence at 6 months after resection.

(limited mesenteric resection).

DETAILED DESCRIPTION:
The current standard of care for ileocolic Crohn's disease (CD) is a limited mesenteric resection. There is growing, but still limited, evidence that extended mesenteric excision during ileocolic resection is beneficial in decreasing disease recurrence. We propose a prospective multicenter cohort study to better understand the role of extended mesenteric excision in ileocolic CD and how it affects disease recurrence. The primary outcome of this study will be the rate of endoscopic recurrence at 6 months in patients undergoing first-time resection for ileocolic CD. Secondary outcomes will include endoscopic recurrence at 18 months and rates of recurrence requiring surgery by 2 years. These outcomes will be compared to historical controls (limited mesenteric resection). Our hypothesis is that patients receiving extended mesenteric ileocolic resection will have reduced endoscopic recurrence at 6 months after resection. As seen in previous studies, advanced mesenteric and mucosal disease predicts increased surgical recurrence.

ELIGIBILITY:
Inclusion Criteria:

adults >18 years old diagnosis of CD limited to the distal ileum/ileocolic region no previous ileocolic resection all forms of CD presentation will be included - stricturing, fistulizing, perforating etc.

Exclusion Criteria:

previous ileocolic resection other sites of CD intraabdominal sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-09-27 (Estimated); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
Endoscopic recurrence at 6 months | 6 months
  Endoscopic recurrence after extended mesenteric ileocolic resection

SECONDARY OUTCOMES:
Endoscopic recurrence at 18 months | 18 months
  Endoscopic recurrence will be evaluated by the endoscopist and will be evaluated according to the Rutgeert's score
Rates of recurrence requiring surgery by 2 years | 24 months
  Surgical recurrence after extended mesenteric ileocolic resection
Post-operative complications | 30 days
  Post-operative complications including: wound infections, anastomotic leak, intra-abdominal abscess, venous-thromboembolic complications, and primary ileus within 30 days of the first resection.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec